CLINICAL TRIAL: NCT06076421
Title: Do Evidence-based Fact Boxes Improve Informed Decision-making About COVID-19 and Influenza Vaccination in More and Less Disadvantaged Groups Equally? - Study Protocol for a Multi-center Cluster RCT in Health and Social Care in Germany
Brief Title: Equity Evaluation of Fact Boxes on Informed COVID-19 and Influenza Vaccination Decisions - Study Protocol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harding Center for Risk Literacy (Other)
Responsible Party: Principal Investigator, Felix G. Rebitschek, Head Research Scientist and CEO, Harding Center for Risk Literacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 57/2022
Record Dates: First submitted 2023-09-29; First posted 2023-10-10 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Influenza
Keywords: health inequity; informed decision making; fact box; evidence-based health information; risk communication
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Intervention Model Description: Cluster randomised cross-sectional controlled trial with a 2x2-design with the between-subjects factors: format (usual care plus evidence-based fact box vs. usual care), health educator (cluster unit medical practice vs. cluster unit outreach work settings) taking into account various factors of disadvantage (e.g., low education).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evidence-based fact box on COVID-19 or influenza (intervention) (Experimental): Health educators (HE) will receive a flyer with a brief description of the study, a Quick Response-code (QR-code) and a link to an online survey, including either a fact box as tabular format or a visualization on the reverse side about COVID-19 or the flu vaccine to distribute to potential study participants. HE are free to decide if and how to use the fact boxes: whether during, before or after vaccination education, and who to target.
  Participants who receive the flyer from their HE can decide on their own to participate in the study by using the QR-code or link on the flyer.
  Interventions: Other: Fact box
- Usual education/care (No Intervention): Study participants whose HE will be randomised to the control will receive the same flyer but without a fact box on the reverse side.

INTERVENTIONS:
Other: Fact box — Fact boxes provide a tabular or graphical overview of the benefits and harms of the COVID-19 or influenza vaccination through transparent risk communication. The fact boxes are available for two different age groups each: COVID-19 vaccination for people aged 18 to 59 and over 60, influenza vaccination for people aged 16 to 64 and over 65 in Arabic, German, Russian and Turkish.
  Arms: Evidence-based fact box on COVID-19 or influenza (intervention)

SUMMARY:
The study aims to evaluate whether evidence-based fact boxes on COVID-19 and influenza vaccination contribute to the decision making of laypeople from different social backgrounds in different educational settings (e.g. medical practices, outreach work). Furthermore, the study will investigate whether evidence-based fact boxes can contribute to more equitable health care by improving shared decision-making.

DETAILED DESCRIPTION:
Background

Evidence-based health information (EBHI) and decision aids (DA) are key components for improving health care by enabling more people to make informed decisions. However, despite their overall effectiveness, there is a risk that only certain groups of the population will benefit from them. Because although they are target group oriented, the factors that lead to inequality in terms of shared and informed decision-making have not yet been sufficiently taken into account in their development process. For example, there are many patient-oriented materials written at an advanced level, which makes the materials less accessible to people with reading difficulties, lower education, health literacy or socioeconomic status (SES).

Evidence-based fact boxes have been shown to support informed decision-making. However, few studies have analysed how the boxes support decision-making in different social groups. Further, it is unclear whether fact boxes promote informed and shared decision making equally when implemented by health educators (HE) in different settings. Hence, there is a risk that fact boxes will only help less disadvantaged people to make informed health decisions.

Objective

In a Multi-center, cluster-randomised, cross-sectional study, the effectiveness of evidence-based fact boxes (intervention) compared with usual health education/care (control) on outcomes relevant to the decision to vaccinate will be investigated in people from different backgrounds in Germany.

Fact boxes on COVID-19 and influenza vaccination have been adapted in several steps to meet the information needs and requirements of the population. This included feedback from various public health stakeholders on a COVID-19 fact box implemented in Germany in January 2021 by a national Public Health institute, the identification of information needs and requirements of the population in Germany based on secondary data analyses, and testing of COVID-19 fact boxes in pre-studies in population-wide surveys with N=1,942 to N=6,056 respondents in Germany. The data basis and individual studies have been described in detail elsewhere.

The Influenza vaccination fact box was updated in 2021 based on current evidence and is available on the Harding Center website for older people (65 years and older) and for people aged 16 to 65. During cognitive interviews, simplified COVID-19 and Influenza vaccination fact boxes were first piloted with German-speaking laypeople and adapted based on their feedback. Visualized COVID-19 fact boxes were also piloted with Arabic-, Turkish- and Russian-speaking laypeople from disadvantaged neighbourhoods in Berlin. A visualized flu fact box is currently being piloted by the University of Erfurt with German-speaking lay people.

Main research question

Do disadvantaged people benefit to the same extent as non-disadvantaged people in terms of informed and shared decision-making from receiving COVID-19 and influenza vaccination fact boxes as opposed to standard vaccination communication in medical practices and outreach work (field settings)?

Research questions (RQ) and main hypotheses (HYP)

RQ1 Is the use of fact boxes more effective than standard vaccine communication (control condition) in the field?

Primary HYP

1. Compared to standard vaccine communication, fact boxes will lead to higher vaccination knowledge.
2. Compared to standard vaccine communication, fact boxes will lead to more vaccination intentions that are in line with attitudes and vaccination knowledge (informed vaccination intentions; operationalised based on the multidimensional construct of informed choice by Marteau et al. 2001).

Secondary HYP

1. Compared to standard vaccine communication, fact boxes will improve risk perception.
2. Compared to standard vaccine communication, fact boxes will increase patient involvement in medical decision making.
3. Compared to standard vaccine communication, fact boxes will decrease decisional conflict.

RQ2 Are fact boxes as effective for people with disadvantaging factors as for those without factors associated with disadvantages?

Primary HYP

Compared to standard vaccine communication, fact boxes will lead to a greater alignment of knowledge, informed vaccination intentions, and accuracy of risk perception between:

1. People with low and high education through fact boxes compared to usual care.
2. People with problematic or inadequate and excellent or sufficient level of health literacy through fact boxes compared to usual care.
3. Non-native (Arabic, Turkish and Russian speaking participants, only with low German skills) and native German speakers (including non-native speakers with high German skills), because the investigators not only provide information in the native language, but also tested it with these target groups.
4. People with low and high reading literacy in different languages, because fact boxes are a complexity-reduced format of health information and the investigators tried to address accessibility through pilot testing with different groups.

RQ3 Does the use of fact boxes in outreach work promote more shared and informed decision-making than in regular health care settings?

HYP

a) Compared to standard vaccine communication fact boxes will more likely lead to more informed vaccination intentions and shared decisions in outreach work than in regular health care settings.

Explorative analyses

1. The investigators will analyse the effect of fact boxes on knowledge, vaccination intentions, accuracy of risk perception between people with low and medium or high SSS through fact boxes compared to usual care.
2. The investigators will analyse the effect of fact boxes on vaccination intentions, knowledge, risk perception, patient involvement, and decisional conflict among people with migration-related indicators (e.g., residential status, length of stay in Germany) compared to usual care, controlling for other factors describing the social situation (e.g., education, health literacy).

ELIGIBILITY:
Inclusion Criteria:

* Adults of legal age with current residence in Germany and who speak Arabic, German, Russian, Turkish
* People who are currently facing a decision about COVID-19 or influenza vaccination for themselves or a family member (e.g. caring relatives)
* Informed online consent

Exclusion Criteria:

* Language other than Arabic, German, Russian, Turkish
* People without a current vaccination decision
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Knowledge | at T1 (initial survey; study period: 3-6 month)
  10 items: five items on basic knowledge of the disease (e.g. how is Corona or the flu contracted and what are the possible baseline risks) and uncertainty (e.g. quality of evidence), each with 4 possible answers, of which only one is correct. A further five questions that can only be answered through the fact box, including one question on the benefits of vaccination gist and three questions on the benefits and harms of vaccination verbatim. Responses will be graded according to the best available evidence in July 2023.
Informed vaccination intention | at T1 (initial survey; study period: 3-6 month)
  Based on vaccination knowledge, a person's attitudes and vaccination intentions.
  Knowledge will be measured as described above. Attitudes will be measured using an 11-point Likert scale that captures the personal assessment of the balance between the potential benefits and risks of the respective vaccine. Vaccination intention will be measured by asking whether participants would have themselves or their relatives vaccinated at the next opportunity, on a scale of 1-5 (Definitely yes, probably yes, probably not, definitely not, I cannot yet say / am still undecided).

SECONDARY OUTCOMES:
Risk perception | at T1 (initial survey; study period: 3-6 month)
  Based on a frequency format (Please imagine 10 people like yourself: How many of them will be re-infected with COVID-19 after a previous coronavirus infection if they come into contact with a person who is infected with the coronavirus variant XBB.1.5?; How many will contract influenza in a year if the virus is widespread?): Correct responses (reflected the best available evidence, which can be found in the fact boxes together with the medical references.
Decisional conflict | at T1 (initial survey; study period: 3-6 month)
  The 4-item SURE (Sure of myself; Understand information; Risk-benefit ratio; Encouragement) screening test will be used (if yes: 1, if no: 0; a score of < 4 is a positive result for decisional conflict)
Patient involvement in decision making | at T1 (initial survey; study period: 3-6 month)
  Measured with the 9-item Shared Decision Making Questionnaire (SDM-Q-9). The instrument contains nine statements which are rated on a six-point Likert scale (from 0 'completely disagree' to 5 'completely agree').

OTHER OUTCOMES:
Health literacy | at T1 (initial survey; study period: 3-6 month)
  Measured by using the established and validated 12-item Health Literacy Survey Questionnaire (HLS19-Q12), a short form questionnaire of the 47-item Health Literacy Survey Questionnaire (HLS19-Q47) for measuring comprehensive, general health literacy (HL) in general adult populations. After an introductory statement about handling health information, respondents are asked to choose one of four response categories to the 12 questions about how easy or difficult tasks related to handling health information are (with 4 'very easy', 3 'easy', 2 'difficult', 1 'very difficult').
Subjective socioeconomic status | at T1 (initial survey; study period: 3-6 month)
  Will be assessed by using the MacArthur Scale of Subjective Social status (SSS), which measures the subjective perception of social position within society on a 10-point scale (with SSS low: 1-4, middle: 5-6, high: 7-10).

CONTACTS AND LOCATIONS:
Overall Officials: Christin Ellermann, MSc, Principal Investigator — Harding Center for Risk Literacy; Felix G. Rebitschek, Dr., Principal Investigator — Harding Center for Risk Literacy
Locations (1):
- Harding Center for Risk Literacy, Faculty of Health Sciences Brandenburg, University of Potsdam, Potsdam, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
All relevant data will be provided in the manuscript and supporting information or made available in a public repository after completion of the study.
Time Frame: After completion of the study.
Access Criteria: All relevant data will be provided in the manuscript and supporting information or made available in a public repository (e.g., OSF) after completion of the study.

REFERENCES:
- [Background] Adler NE, Epel ES, Castellazzo G, Ickovics JR. Relationship of subjective and objective social status with psychological and physiological functioning: preliminary data in healthy white women. Health Psychol. 2000 Nov;19(6):586-92. doi: 10.1037//0278-6133.19.6.586. PMID 11129362
- [Background] Pelikan JM, Link T, Strassmayr C, Waldherr K, Alfers T, Boggild H, Griebler R, Lopatina M, Miksova D, Nielsen MG, Peer S, Vrdelja M; HLS19 Consortium of the WHO Action Network M-POHL. Measuring Comprehensive, General Health Literacy in the General Adult Population: The Development and Validation of the HLS19-Q12 Instrument in Seventeen Countries. Int J Environ Res Public Health. 2022 Oct 29;19(21):14129. doi: 10.3390/ijerph192114129. PMID 36361025
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Legare F, Kearing S, Clay K, Gagnon S, D'Amours D, Rousseau M, O'Connor A. Are you SURE?: Assessing patient decisional conflict with a 4-item screening test. Can Fam Physician. 2010 Aug;56(8):e308-14. PMID 20705870
- [Background] Rebitschek FG, Ellermann C, Jenny MA, Siegel NA, Spinner C, Wagner GG. Fact boxes that inform individual decisions may contribute to a more positive evaluation of COVID-19 vaccinations at the population level. PLoS One. 2022 Sep 12;17(9):e0274186. doi: 10.1371/journal.pone.0274186. eCollection 2022. PMID 36095020
- [Background] Marteau TM, Dormandy E, Michie S. A measure of informed choice. Health Expect. 2001 Jun;4(2):99-108. doi: 10.1046/j.1369-6513.2001.00140.x. PMID 11359540
- [Background] Durand MA, Yen RW, O'Malley AJ, Schubbe D, Politi MC, Saunders CH, Dhage S, Rosenkranz K, Margenthaler J, Tosteson ANA, Crayton E, Jackson S, Bradley A, Walling L, Marx CM, Volk RJ, Sepucha K, Ozanne E, Percac-Lima S, Bergin E, Goodwin C, Miller C, Harris C, Barth RJ Jr, Aft R, Feldman S, Cyr AE, Angeles CV, Jiang S, Elwyn G. What matters most: Randomized controlled trial of breast cancer surgery conversation aids across socioeconomic strata. Cancer. 2021 Feb 1;127(3):422-436. doi: 10.1002/cncr.33248. Epub 2020 Nov 10. PMID 33170506
- [Background] Miller DP Jr, Spangler JG, Case LD, Goff DC Jr, Singh S, Pignone MP. Effectiveness of a web-based colorectal cancer screening patient decision aid: a randomized controlled trial in a mixed-literacy population. Am J Prev Med. 2011 Jun;40(6):608-15. doi: 10.1016/j.amepre.2011.02.019. PMID 21565651
- [Derived] Ellermann C, Savaskan N, Rebitschek FG. Do summaries of evidence enable informed decision-making about COVID-19 and influenza vaccination equitably across more and less disadvantaged groups? Study protocol for a multi-centre cluster randomised controlled trial of 'fact boxes' in health and social care in Germany. BMJ Open. 2024 Nov 1;14(10):e083515. doi: 10.1136/bmjopen-2023-083515. PMID 39486820